CLINICAL TRIAL: NCT00862953
Title: The Lifestyle, OverWeight, Energy Restriction Study
Brief Title: Study to Assess the Effects of High Protein Diet in Obesity, the LOWER Study
Acronym: LOWER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BWO08-002
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Obesity
Keywords: low carbohydrate; high protein diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal protein normal carbohydrate (Active Comparator): Normal protein normal carbohydrate calory restricted nutrition
  Interventions: Dietary Supplement: Normal protein energy-restricted
- Normal protein low carbohydrates (Experimental): Normal protein low carbohydrate energy-restricted diet
  Interventions: Dietary Supplement: Normal protein energy-restricted
- High protein normal carbohydrates (Experimental): High protein normal carbohydrates
  Interventions: Dietary Supplement: High protein energy-restricted
- High protein low carbohydrate (Experimental): High protein low carbohydrate nutrition
  Interventions: Dietary Supplement: High protein energy-restricted

INTERVENTIONS:
Dietary Supplement: Normal protein energy-restricted — Normal protein diet energy restricted
  Arms: Normal protein low carbohydrates; Normal protein normal carbohydrate
Dietary Supplement: High protein energy-restricted — High protein diet, with either low or normal carbohydrate content
  Arms: High protein low carbohydrate; High protein normal carbohydrates

SUMMARY:
This program is carried out in a dedicated outpatient-clinic in the city of Hengelo for the evaluation and treatment of subjects with obesity. The program puts emphasis on intervention with appropriate diet and physical exercise, and supports the patients in achieving long-term behaviour changes. Interventions which are compared are normal vs high protein/low carb diets.

DETAILED DESCRIPTION:
Assessment focuses on the effect of the specific diets on weight reduction after 3 months, and weight maintenance after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Obesity with BMI > 27 kg/m2

Exclusion Criteria:

* Recent loss of body weight (>10%)
* Underlying malignancy, HIV infection, psychiatric disease
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Body weight | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: F NR Van Berkum, MD PhD, Study Director — Previtas Hengelo
Locations (1):
- Hospital Hengelo, Hengelo, Netherlands